CLINICAL TRIAL: NCT01148355
Title: Effects of Smoking Cues on Tobacco Craving Responses and the Reinforcing Efficacy of Cigarettes in Adolescent Smokers
Status: Completed | Type: Observational
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999908435; 08-DA-N435
Record Dates: First submitted 2010-06-19; First posted 2010-06-22 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-01-14

CONDITIONS: Nicotine Dependence
Keywords: Craving; Moods; Adolescents; Nicotine; Reinforcement
MeSH Terms: conditions — Tobacco Use Disorder

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

* Multiple social, psychological, and environmental factors contribute to adolescents' use of cigarettes. Environmental smoking cues have been shown to play an important role in the maintenance of nicotine addiction and in relapse to smoking. However, few studies have examined craving and cue-reactivity in adolescent smokers, even though craving appears to contribute to ongoing smoking and relapse in this age group.
* Another factor central to addiction is the rewarding effect of drugs, or the interaction between the person, the drug, and the environmental setting. However, more research is needed on whether environmental cues lead to increased smoking in adolescents.

Objectives:

- To determine the effects of smoking versus neutral cues in adolescents who smoke on (1) craving, mood, and autonomic responsivity and (2) the relative reinforcing efficacy of tobacco cigarettes.

Eligibility:

- Adolescents 12 to 17 years of age who are current smokers (at least five cigarettes per day for the past 6 months).

Design:

* This study will involve three study visits. Participants will be allowed to smoke before all study sessions and will give a breath carbon monoxide (CO) sample before all sessions. Participants must not use any illicit drugs or alcohol 24 hours before sessions.
* Visit 1 (baseline session): Participants will provide a urine sample and will be familiarized with the study room and session design.
* Visits 2 and 3: Participants will be connected to physiological recording devices to measure heart rate, perspiration, and other physical responses. After baseline readings, participants will be exposed to smoking cues at one experimental session and to neutral cues at the other experimental session.
* Before, during, and after cue presentation, participants will complete self-report measures of mood and craving and have physiological measures taken. They will then be re-exposed to smoking or neutral cues and engage in a self-administration procedure to examine the effect of cues on the reinforcing efficacy of cigarettes.

DETAILED DESCRIPTION:
Objective:

To determine the effects of smoking versus neutral cues in adolescents who smoke on 1) craving, mood, and autonomic responsivity and 2) the relative reinforcing efficacy of tobacco cigarettes.

Study population:

25 adolescents who smoke at least 5 cigarettes per day.

Design:

Comparison-controlled, within-subjects design.

Outcome Measures:

During cue trials, primary measures include craving (TCQ-SF, VAS), mood (mood form, VAS), and autonomic (heart rate, blood pressure, skin conductance) responsivity. During self-administration trials, primary measures include breakpoint (final ratio completed), total number of responses, and number of cigarette puffs earned and taken. Secondary measures include baseline smoking history, mood, tobacco craving, smoking expectancies, nicotine dependence, and urinary cotinine and 3-hydroxycotinine.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. 13-17 year old males and females
  2. smoking at least 5 cigarettes per day for at least 6 months
  3. urinary cotinine level greater than or equal to 100 ng/ml (NicAlert(Registered Trademark) reading greater than or equal to 3)
  4. medically and psychologically healthy as determined by screening criteria.

EXCLUSION CRITERIA:

1. current interest in reducing or quitting smoking
2. treatment for nicotine dependence in the past 3 months
3. use of nicotine replacement products, bupropion, or varenicline in the past 3 months
4. alcohol and any illicit drug use more than 7 times in the last 14 days
5. current use of any medication that would interfere with the protocol in the opinion of MAI
6. pregnant, nursing, or become pregnant during the study

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 25 (Estimated)
Dates: Start 2008-06-10; Study Completion 2011-01-14

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute on Drug Abuse, Biomedical Research Center (BRC), Baltimore, Maryland, United States

REFERENCES:
- [Background] Bagot KS, Heishman SJ, Moolchan ET. Tobacco craving predicts lapse to smoking among adolescent smokers in cessation treatment. Nicotine Tob Res. 2007 Jun;9(6):647-52. doi: 10.1080/14622200701365178. PMID 17558821
- [Background] Bickel WK, Hughes JR, DeGrandpre RJ, Higgins ST, Rizzuto P. Behavioral economics of drug self-administration. IV. The effects of response requirement on the consumption of and interaction between concurrently available coffee and cigarettes. Psychopharmacology (Berl). 1992;107(2-3):211-6. doi: 10.1007/BF02245139. PMID 1615122
- [Background] Corrigall WA. Nicotine self-administration in animals as a dependence model. Nicotine Tob Res. 1999 Mar;1(1):11-20. doi: 10.1080/14622299050011121. PMID 11072385